CLINICAL TRIAL: NCT04050683
Title: Evaluation of Hemodynamic Parameters Following Transjugular Intrahepatic Portosystemic Shunt (TIPS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Radiological Society of North America (Other)
Responsible Party: Principal Investigator, Eric J. Hohenwalter, MD, Professor of Radiology, Vascular & Interventional Radiology, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO 35079
Record Dates: First submitted 2019-08-07; First posted 2019-08-08 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Refractory Ascites
Keywords: TIPS; Hemodynamic; Ascites; Hepatic; Hydrothorax
MeSH Terms: conditions — Ascites; Hydrothorax

STUDY DESIGN:
Intervention Model Description: All patients undergoing TIPS will have the following hemodynamic measurements obtained: systolic, diastolic and mean RAP; systolic, diastolic and mean right ventricular pressure (RSV). Peak systolic right ventricular (PSRV) pressure will serve as surrogate for pulmonary artery pressure (PAP). There are 2 groups in this project. Subjects will be enrolled in 1 of the 2 groups based on their heart pressure measurements (high or normal). If a subject does not meet criteria for 1 of the 2 groups, they will not be in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study - Transjugular Intrahepatic Portosystemic Shunt (TIPS) (Experimental): Right Atrial Pressure (RAP) ≥ 15mmHg or change in RAP ≥ 10 mmHg or Peak Systolic Right Ventricular (PSRV) Pressure ≥ 46 mmHg
  Interventions: Procedure: Study - Transjugular Intrahepatic Portosystemic Shunt (TIPS)
- Control - Transjugular Intrahepatic Portosystemic Shunt (TIPS) (Active Comparator): Normal hemodynamic parameters
  Interventions: Procedure: Control - Transjugular Intrahepatic Portosystemic Shunt (TIPS)

INTERVENTIONS:
Procedure: Study - Transjugular Intrahepatic Portosystemic Shunt (TIPS) — Prior to and 1-3 days after the TIPS procedure, the following blood tests are done for research purposes: Brain Natriuretic Peptide (BNP); Endothelin-1; Tumor Necrosis Factor-alpha (TNF-a); Endothelial Nitric Oxide Synthase (eNOS). Subjects with abnormal heart pressures during TIPS will have a right heart catheterization (RHC) to monitor heart function, blood flow, and pressures in and around the heart. The subject will be admitted to the Cardiovascular Intensive Care Unit and have a TTE all of which are standard of care. Routine follow-up visits will occur in IR Clinic at 2 Weeks (± 3 days), 4-6 weeks and 4-6 months. Visits will include: blood draws for research related blood tests as listed above; standard of care ultrasound of the abdomen; TTEs; and for at least one year, routine lab testing, imaging, medications, and subject overall condition will be assessed for long term outcomes. Diagnostic RHC will be done as needed per standard of care.
  Other Names: Hemodynamic Measurements; Transthoracic Echocardiogram (TTE); Research Blood Tests
  Arms: Study - Transjugular Intrahepatic Portosystemic Shunt (TIPS)
Procedure: Control - Transjugular Intrahepatic Portosystemic Shunt (TIPS) — Subject's with normal heart pressures who are having elective (planned in advance and not due to an emergency) TIPS due to refractory ascites (fluid build up in the belly that does not go away or comes back shortly after being removed). Prior to and 1-3 days after the TIPS procedure, the following blood tests are done for research purposes: Brain Natriuretic Peptide (BNP); Endothelin-1; Tumor Necrosis Factor-alpha (TNF-a); Endothelial Nitric Oxide Synthase (eNOS). The subject will be admitted to the hospital after TIPS for standard of care monitoring.
  Routine follow-up visits will occur in IR Clinic at 2 Weeks (± 3 days), 4-6 weeks and 4-6 months. Visits will include: blood draws for research related blood tests as listed above; standard of care ultrasound of the abdomen; and for at least one year, routine lab testing, imaging, medications, and subject overall condition will be assessed for long term outcomes.
  Other Names: Hemodynamic Measurements; Research Blood Tests
  Arms: Control - Transjugular Intrahepatic Portosystemic Shunt (TIPS)

SUMMARY:
During a TIPS procedure, a shunt or stent (mesh tube) is passed down the jugular vein (the vein above the collarbone in the neck) using fluoroscopy (real time x-rays) guidance. Then, a stent is inserted between the portal vein (vein that carries blood from the intestines into the liver) to a hepatic vein (vein that carries blood away from the liver back to the heart). This means that blood that would usually gets filtered through the liver is now bypassing the liver and going directly to the heart. Because more blood will be flowing to the heart, the heart needs to be strong enough to handle the extra volume.

This study is being done to determine the impact of the TIPS procedure on cardiac (heart) function by collecting data (heart pressures) during the TIPS procedure. Immediately after TIPS and at standard follow-up time points, labs and transthoracic echocardiograms (TTE or echo) will also be collected.

The device(s) used in this study are neither the intervention studied nor the experimental variable of interest. Devices are commercially available and used, and procedures are performed, in accordance with the institution's standard of care.

DETAILED DESCRIPTION:
The long-term goal of this proposal is to improve survival in patients with end stage liver disease following TIPS placement. Given that the most common indications for TIPS placement are also defining features of decompensated cirrhosis, specifically hemorrhage and refractory ascites, the overall health of this patient population is extraordinarily complex. One notable circulatory impact of cirrhosis is the increase in total blood volume in concert with a disproportionate increase in splanchnic blood volume. Therefore, at the time of TIPS placement, a patient may experience a marked increase in central blood volume that may lead to cardiac dysfunction. Considering that a central feature of cirrhotic cardiomyopathy is attenuated response to stress, it is conceivable that some perioperative cardiovascular complications could be attributed to the patient's baseline health rather than an isolated effect of the procedure alone. By instituting measures to identify patients that may be at increased risk for an adverse outcome, this proposal hopes to offer a new paradigm for managing TIPS patients in the acute postoperative setting. Therefore, the purpose of this study is to derive better correlates between non-invasive and invasive measurements of cardiac function.

ELIGIBILITY:
OVERALL INCLUSION

* ≥ 18 years
* Patients with indications as established by the ACR-SIR-SPR practice parameters::

  * prophylaxis against recurrent variceal bleed in high-risk patients
  * portal hypertensive gastropathy or intestine-opathy
  * refractory ascites
  * hepatic hydrothorax
  * hepatopulmonary syndrome
  * hepatorenal syndrome
  * decompression of portosystemic collaterals prior to abdominal surgical procedures
* Technically successful creation of a TIPS shunt, defined as creation of a portosystemic shunt with post TIPS creation portosystemic gradient of ≤ 12 mmHg

STUDY ARM INCLUSION:

• All patients undergoing elective TIPS who meet at least one of the criteria:

* Right atrial pressure (RAP) ≥ 15mm Hg; OR
* Change in RAP ≥ 10mm Hg; OR
* Peak systolic velocity ratio (PSRV) pressure ≥ 46mm Hg

CONTROL ARM INCLUSION:

• Patients undergoing elective TIPS for control of refractory ascites who do not meet at least one of the criteria outlined above for the study arm.

Historical controls: we will use data collected form our own recent institutional review.

EXCLUSION All patients who do not exhibit alterations in invasive RAP or PRVS measurements as listed in Inclusion Criteria and do not meet criteria for participation as a control subject (i.e. are not undergoing elective TIPS for control of refractory ascites).

Admitted for GI bleed.

Budd-Chiari syndrome.

TIPS in setting of mesenteric vein thrombosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Cardiac related events | from insertion of TIPS to 1 year post TIPS
  any cardiac event to include, heart failure, heart attack, pulmonary hypertension

SECONDARY OUTCOMES:
Clinical success | 6 months after TIPS placement
  No further need for paracentesis or thoracentesis at 6 months
Overall survival | all patients will be followed for 1 year after TIPS placement
  evaluation of overall survival from time of TIPS placement to death
Complications | from insertion of TIPS to 1 year post TIPS
  Any peri or post procedural TIPS related events including liver failure, need for re-intervention, etc.
TIPS patency | from insertion of TIPS to 1 year post TIPS
  evaluation of how long the TIPS remains patent without need for further intervention

OTHER OUTCOMES:
Correlation of cardiac events with laboratory values | labs will be obtained at baseline and post TIPS at 1-3 days, 2 weeks +/- 3 days, 4-6 weeks, and 4-6 months
  correlations will be made between outcome BNP, TNF-a, eNOS, endothelin-1

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Hohenwalter, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants must have agreed to banking of biosamples. Identified individual participant data for all primary and secondary outcome measures will be made available. Also, left-over research related blood samples will be retained in an IRB approved bank.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: During and after (indefinitely) study participation.
Access Criteria: Participants must have signed the biosample bank consent.

REFERENCES:
- [Background] Strizhakov AN, Lebedev VA. [The current approaches to choosing a rational procedure for the pregnancy and labor management of women with a scar on the uterus]. Akush Ginekol (Mosk). 1991 Feb;(2):8-13. No abstract available. Russian. PMID 1862861
- [Background] ACR-SIR-SPR Practice Parameter for the Creation of a Transjugular Intrahepatic Portosystemic Shunt (TIPS). :25.
- [Background] Ascha M, Abuqayyas S, Hanouneh I, Alkukhun L, Sands M, Dweik RA, Tonelli AR. Predictors of mortality after transjugular portosystemic shunt. World J Hepatol. 2016 Apr 18;8(11):520-9. doi: 10.4254/wjh.v8.i11.520. PMID 27099653
- [Background] Parvinian A, Bui JT, Knuttinen MG, Minocha J, Gaba RC. Right atrial pressure may impact early survival of patients undergoing transjugular intrahepatic portosystemic shunt creation. Ann Hepatol. 2014 Jul-Aug;13(4):411-9. PMID 24927612
- [Background] Kiszka-Kanowitz M, Henriksen JH, Moller S, Bendtsen F. Blood volume distribution in patients with cirrhosis: aspects of the dual-head gamma-camera technique. J Hepatol. 2001 Nov;35(5):605-12. doi: 10.1016/s0168-8278(01)00175-1. PMID 11690706
- [Background] Xu J, Murphy SL, Kochanek KD, Bastian B, Arias E. Deaths: Final Data for 2016. Natl Vital Stat Rep. 2018 Jul;67(5):1-76. PMID 30248015
- [Background] Marcellin P, Kutala BK. Liver diseases: A major, neglected global public health problem requiring urgent actions and large-scale screening. Liver Int. 2018 Feb;38 Suppl 1:2-6. doi: 10.1111/liv.13682. PMID 29427496
- [Background] Barger IA, Le Jambre LF, Georgi JR, Davies HI. Regulation of Haemonchus contortus populations in sheep exposed to continuous infection. Int J Parasitol. 1985 Oct;15(5):529-33. doi: 10.1016/0020-7519(85)90049-9. No abstract available. PMID 4066146
- [Background] Ruiz-del-Arbol L, Serradilla R. Cirrhotic cardiomyopathy. World J Gastroenterol. 2015 Nov 7;21(41):11502-21. doi: 10.3748/wjg.v21.i41.11502. PMID 26556983
- [Background] Luo B, Liu L, Tang L, Zhang J, Ling Y, Fallon MB. ET-1 and TNF-alpha in HPS: analysis in prehepatic portal hypertension and biliary and nonbiliary cirrhosis in rats. Am J Physiol Gastrointest Liver Physiol. 2004 Feb;286(2):G294-303. doi: 10.1152/ajpgi.00298.2003. PMID 14715521
- [Background] Tsiakalos A, Hatzis G, Moyssakis I, Karatzaferis A, Ziakas PD, Tzelepis GE. Portopulmonary hypertension and serum endothelin levels in hospitalized patients with cirrhosis. Hepatobiliary Pancreat Dis Int. 2011 Aug;10(4):393-8. doi: 10.1016/s1499-3872(11)60066-0. PMID 21813388
- [Background] Ortiz-Muniz G, Sigel MM. Long-term synthesis of antibody in vitro. Proc Soc Exp Biol Med. 1967 Apr;124(4):1178-82. doi: 10.3181/00379727-124-31957. No abstract available. PMID 6024829
- [Background] Boyer TD, Haskal ZJ; American Association for the Study of Liver Diseases. The Role of Transjugular Intrahepatic Portosystemic Shunt (TIPS) in the Management of Portal Hypertension: update 2009. Hepatology. 2010 Jan;51(1):306. doi: 10.1002/hep.23383. No abstract available. PMID 19902484
- [Background] Hoeper MM, Krowka MJ, Strassburg CP. Portopulmonary hypertension and hepatopulmonary syndrome. Lancet. 2004 May 1;363(9419):1461-8. doi: 10.1016/S0140-6736(04)16107-2. PMID 15121411
- [Background] Ghaferi AA, Birkmeyer JD, Dimick JB. Complications, failure to rescue, and mortality with major inpatient surgery in medicare patients. Ann Surg. 2009 Dec;250(6):1029-34. doi: 10.1097/sla.0b013e3181bef697. PMID 19953723
- [Background] Preston SR, Markar SR, Baker CR, Soon Y, Singh S, Low DE. Impact of a multidisciplinary standardized clinical pathway on perioperative outcomes in patients with oesophageal cancer. Br J Surg. 2013 Jan;100(1):105-12. doi: 10.1002/bjs.8974. Epub 2012 Nov 12. PMID 23161343
- [Background] Sinclair S, James S, Singer M. Intraoperative intravascular volume optimisation and length of hospital stay after repair of proximal femoral fracture: randomised controlled trial. BMJ. 1997 Oct 11;315(7113):909-12. doi: 10.1136/bmj.315.7113.909. PMID 9361539
- [Background] Nevah MI, Kuruvilla AC, Fallon MB. Cardiopulmonary Complications of Cirrhosis. Zakim and Boyer's Hepatology. 7th ed. Philadelphia, PA: Elsevier; 2018 [cited 2018 Dec 22]. p. 281-292.e5.